CLINICAL TRIAL: NCT00647582
Title: Phase II Study of Intra-operative Electron Irradiation and External Beam Irradiation After Lumpectomy in Patients With Stage T1N0M0 or T2N0M0 Breast Cancer
Brief Title: Radiation Therapy During and After Lumpectomy in Treating Women With Stage I or Stage II Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: William Wailing Wong, M.D., Mayo Clinic Cancer Center
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000588774; P30CA015083 (NIH); MCS066 (Other: Mayo Clinic Cancer Center); 1681-02 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2008-03-28; First posted 2008-03-31 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2016-04

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Chemotherapy, Adjuvant; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: adjuvant therapy
Procedure: therapeutic conventional surgery
Radiation: intraoperative radiation therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiation therapy during and after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying the side effects of giving radiation therapy during and after lumpectomy and to see how well it works in treating women with stage I or stage II breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the feasibility and acute tolerability of intraoperative electron radiotherapy (IOERT) and external-beam radiotherapy (EBRT) after lumpectomy in women with stage I or II breast cancer treated with breast conservation therapy.
* To determine the local tumor control and distant tumor control rates in these patients.
* To determine the long-term side effects and cosmetic outcome of IOERT to the tumor bed and EBRT after lumpectomy in these patients.

OUTLINE: Patients undergo standard lumpectomy. Patients with negative lymph nodes undergo intraoperative electron radiotherapy to the tumor bed. Beginning 2-8 weeks after surgery, patients undergo whole breast external beam radiotherapy once daily for 24-27 fractions.

After completion of study treatment, patients are followed periodically for up to 8 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary invasive breast carcinoma, meeting the following criteria:

  * Stage I or II disease (T1-T2, N0, M0)
  * Tumor pathologically determined to be ≤ 5 cm in diameter
  * Single, discrete, well-defined primary tumor
* No multicentric disease and/or diffuse malignant appearing microcalcifications

  * Any microcalcifications must be focal

    * Specimen radiograph is required after lumpectomy to assure removal of all malignant appearing calcifications
* No axillary lymph node involvement

  * Axillary lymph node status can be determined by level I and II lymph node dissection or sentinel lymph node sampling
* Must have pathologically negative surgical margins
* No evidence of metastatic breast cancer
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Menopausal status not specified
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No pre-existing collagen vascular disease except rheumatoid arthritis that does not require immunosuppressive therapy

PRIOR CONCURRENT THERAPY:

* No prior irradiation to the area of planned radiation field
* Concurrent hormone therapy allowed

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2002-10; Primary Completion 2005-06 (Actual); Study Completion 2013-12-21 (Actual)

PRIMARY OUTCOMES:
Feasibility
Acute tolerability
Local tumor control rate
Distant tumor control rate
Long-term side effects
Cosmetic outcome

CONTACTS AND LOCATIONS:
Overall Officials: William W. Wong, MD, Study Chair — Mayo Clinic